CLINICAL TRIAL: NCT06005012
Title: Semaglutide Treatment in the Real-world for Fibrosis Due to NAFLD in Obesity and T2DM
Acronym: SAMARA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRC-2023-1
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Fibrosis, Liver; Type 2 Diabetes Mellitus in Obese; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): 2.4 mg weekly for 52 weekly in a 3 ml PDS290 pen-injector containing Semaglutide 3.0 mg/ml for subcutaneous use
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): 2.4 mg weekly for 52 weekly in a 3 ml PDS290 pen-injector containing 3.0 mg/ml of a placebo solution for subcutaneous use
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide is a glucagon-like peptide 1 receptor agonist (GLP-1 RA) that is FDA-approved for the treatment of obesity (as Wegovy) or T2DM (as Ozempic).
  Arms: Semaglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Conduct a community intervention study that will 1) validate a screening approach to identify patients at risk for advanced NAFLD in the obese or T2DM population, and 2) test whether semaglutide treatment is effective for the management of significant fibrosis due to NAFLD in high-risk patients.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) affects approximately 25-30% of the global population and is projected to become the leading cause of liver transplantation in the United States by 2030. Development of efficient screening strategies for the identification and treatment of individuals who are at greatest risk for advanced disease in this population is an urgent and unmet medical need. Type 2 diabetes mellitus (T2DM) and obesity are critical risk factors for advanced NAFLD. In a prospective cross-sectional study of patients with type 2 diabetes, we screened 524 participants (50-80 years old) with type 2 diabetes mellitus for the presence of NAFLD and observed relative prevalences of 70% for steatosis and 15% for advanced fibrosis. The presence of obesity in this population further increased the odds of advanced fibrosis. These findings suggest that screening populations of individuals with obesity or T2DM may be an effective strategy for identifying high-risk patients with NAFLD. Semaglutide is a glucagon-like peptide 1 receptor agonist (GLP-1 RA) that is FDA-approved for the treatment of obesity (as Wegovy) or T2DM (as Ozempic), conditions that are considered major risk factors for advanced fibrosis in the NAFLD population. It is unclear, however, whether semaglutide is effective for treatment of fibrosis due to NAFLD in these populations. Here, the investigators propose to conduct a community intervention study that will 1) validate a screening approach to identify patients at risk for advanced NAFLD in the obese or T2DM population, and 2) test whether semaglutide treatment is effective for the management of significant fibrosis due to NAFLD in high-risk patients.

ELIGIBILITY:
Inclusion criteria:

1. Adult, age ≥ 40 and < 80 years
2. Participant must meet at least one of following sets of conditions:

   1. BMI ≥ 27 kg/m² OR
   2. BMI ≥ 25 kg/m² AND presence of i) pre-diabetes (HbA1C ≥ 5.7) or ii) type 2 diabetes mellitus (T2DM), as defined by the American Diabetes Association (ADA) clinical practice recommendations.

   The ADA definition of T2DM is applicable if one of the following criteria is met:
   * Presence of diabetes symptoms (polyuria, polydipsia, polyphagia, increased fatigue, weight loss, blurred vision) and casual plasma glucose ≥ 200 mg/dL (11.1 mmol/L)
   * Fasting plasma glucose (FPG) ≥ 126 mg/dl (7.0 mmol/L)
   * Plasma glucose ≥ 200 mg/dL (11.1 mmol/L) during a 75-g oral glucose tolerance test (OGTT)⁶⁸. If any of the above test results occur, testing should be repeated on a different day to confirm the diagnosis.

   OR

   • Hemoglobin A1C (HbA1C) ≥ 6.5% ⁶⁹.
3. FAST score ≥ 0.5 and VCTE ≥ 8.0 kPa; FAST score threshold based on data from MAESTRO-NASH trial⁴²; VCTE cutpoint based on AASLD guidelines for identification of patients with significant fibrosis risk.
4. Participants without a VCTE assessment in their medical record may qualify for the study if they have a FIB-4 ≥ 1.0, which is a cutpoint based on observations of patients with T2DM in Ajmera et al³⁰, and VCTE ≥ 8.0 kPa.
5. The subject is fully informed and willing and able to perform all the procedures specified in the protocol and has signed a written informed consent to participate

Exclusion criteria:

1. Presence of regular and/or excessive use of alcohol, defined as > 30 g/day for males and > 20 g/day for females, for a period longer than 2 years at any time in the last 10 years
2. Evidence of cirrhosis or previously known cirrhosis, based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
3. VCTE ≥ 20 kPa
4. Platelet count ≤ 140,000 per Ml
5. Albumin < 3.6 g/dL
6. INR > 1.35, unless on coumadin for another indication
7. Serum creatinine > 2.0 mg/dL
8. eGFR < 30 mL/min/1.73 m² as defined according to the CKDEPI creatinine equation⁷⁰
9. Use of other weight loss medications, including GLP1RA within the last 90 days
10. Greater than 10% weight loss in the prior six months
11. Known or suspected hypersensitivity to GLP1RA medications including semaglutide
12. History of bariatric surgery within the past 5 years or expected bariatric surgery
13. Evidence of other causes of chronic liver disease including:

    1. Hepatitis B, as defined as presence of hepatitis B surface antigen (HBsAg).
    2. Previous or current infection with Hepatitis C, as defined by presence of hepatitis C virus Ab in serum (anti-HCV Ab).
    3. Autoimmune hepatitis, as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
    4. Autoimmune cholestatic liver disorders, as defined by elevation of alkaline phosphatase and anti- mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
    5. Wilson disease, as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease deficiency, as defined by alpha-1-antitrypsin phenotype and liver histology consistent with alpha-1-antitrypsin deficiency.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in fibrosis due to NAFLD | 52 weeks
  Change in fibrosis due to Nonalcoholic fatty liver disease (NAFLD), as measured by change in FAST Score, which combines FibroScan results with aspartate aminotransferase (AST).

SECONDARY OUTCOMES:
Change in liver stiffness | 52 weeks
  Change in liver stiffness, as measured by change in Vibration-Controlled Transient Elastography
Change in steatosis | 52 weeks
  Change in steatosis, as measure by a change in proton density fat fraction or controlled attenuation parameter
Change in ALT | 52 weeks
  Change in ALT, as measured by a change in patients with ALT >= 30 U/L at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States